CLINICAL TRIAL: NCT01477957
Title: The Effect of Bariatric Surgery on Insulin Sensitivity and Energy Metabolism in Obesity Grade 2 -3
Brief Title: The Effect of Bariatric Surgery on Insulin Sensitivity and Energy Metabolism
Acronym: BARIA-DDZ
Status: Recruiting | Type: Observational
Sponsor: German Diabetes Center (Other)
Collaborators: Dep.of General-, Visceral- and Pediatric Surgery, HHU, Duesseldorf, Germany (Unknown); Dep.for Metabolic Diseases, HHU, Duesseldorf, Germany (Unknown); Hospital Neuwerk, Mönchengladbach, Duesseldorf, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: BARIA-DDZ
Record Dates: First submitted 2011-11-13; First posted 2011-11-23 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: weight loss after bariatric surgery; Insulin sensitivity; insulin resistance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Surgical Procedures, Operative; Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Surgery: bariatric surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — biliopancreatic diversion, gastric banding, gastric sleeve resection
  Other Names: bariatric surgery

SUMMARY:
The purpose of this study is:

1. To explore to what extent insulin sensitivity, energy metabolism and ectopic lipid storage can be improved by bariatric surgery
2. To explore to what extent hepatic and muscular disorders of energy metabolism occur in patients with obesity (degree 2-3)
3. To explore whether the steato liver occurring in patients with obesity (degree 2-3) is associated with the degree of liver inflammation

DETAILED DESCRIPTION:
Insulin resistance strongly relates to ectopic lipid deposition in skeletal muscle and the liver, which correlate with insulin resistance. Lipid metabolites accumulating in skeletal muscle and the liver are thought to impair insulin signalling and thereby reduce glucose uptake and glycogen storage. Insulin resistant humans frequently present with decreased mitochondrial function in skeletal muscle which might contribute to lipid accumulation and the development of insulin resistance. Metabolic dysfunction-associated steatotic liver disease comprises steatosis, steatohepatitis and cirrhosis. MASLD correlates with insulin resistance, increased risk for cardiovascular diseases and type 2 diabetes. The mechanisms leading from steatosis to steatohepatitis and insulin resistance in the liver are yet unclear. Bariatric surgery aims at profound reduction of body weight. Also, it frequently and rapidly leads to normalization of glucose tolerance even before the onset of body weight reduction. The underlying mechanisms are yet unclear. In this study we aim to explore the mechanisms underlying the onset of insulin resistance and steatohepatitis in patients with steatosis and to identify the mechanisms leading to improved glucose tolerance in humans after bariatric surgery. We test the following hypotheses: increased lipid availability leads to (i) increased lipid oxidation and oxidative stress (ii) accumulation of lipid metabolites that impair insulin signalling (iii) bariatric surgery improves insulin sensitivity by increasing lipid oxidation.

This study will contribute to the understanding of MASLD and will help to identify new targets for the therapy of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 20 years- ≤ 70 years
* BMI 20- 25 kg/m 2 normal- weight group
* BMI 35- 39,9 kg/m 2 (Obesity grade 2)
* BMI >40 kg/m 2 (Obesity grade 3)

Exclusion Criteria:

* Acute illness 2 weeks before start of examination
* Autoimmune or Immune disorder diseases (Leukozyten < 5000/µl
* Renal insufficiency (Kreatin > 1,5 mg/dl)
* Heart disease, condition after heart attack
* Anemia (Hb <12g/l, controlled before every day of examination) or blood donations 4weeks before examination.
* Participation in another trial within the last 2 weeks
* Pharmacological- immunotherapy (Cortisol, Antihistaminika, ASS)
* Thyroid disorders
* Glitazone Therapy
* Pregnancy, Lactation, Menstruation
* Smoking cigarettes, Alcohol- and drug abuse
* Psychiatric disorders
* Risk for/ or diagnosed HIV/ AIDS or Hepatitis B/C
* Liver disease, which are not caused by non- alcoholic steato- hepatitis
* Working on night shifts or irregular rhythm of night- day
* Impaired wound healing or clotting disorders
* Allergic reaction to local anesthetics
* Malignant cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with obesity and various stages of MASLD, that qualify for bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-09; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Energy metabolism | 5 years
  whole body substrate oxidation, ex vivo mitochondrial function via measurement of high resolution respirometry and in vivo mitochondrial function via measurement of ATP production

SECONDARY OUTCOMES:
weight loss | 5 years
  body weight and body composition before and after bariatric surgery
Insulin sensitivity | 5 years
  Whole body glucose uptake and endogenous glucose production as measure of skeletal muscle and hepatic insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Koliaki C, Szendroedi J, Kaul K, Jelenik T, Nowotny P, Jankowiak F, Herder C, Carstensen M, Krausch M, Knoefel WT, Schlensak M, Roden M. Adaptation of hepatic mitochondrial function in humans with non-alcoholic fatty liver is lost in steatohepatitis. Cell Metab. 2015 May 5;21(5):739-46. doi: 10.1016/j.cmet.2015.04.004. PMID 25955209
- [Derived] Kahl S, Strassburger K, Pacini G, Trinks N, Pafili K, Mastrototaro L, Dewidar B, Sarabhai T, Trenkamp S, Esposito I, Schlensak M, Granderath FA, Roden M. Dysglycemia and liver lipid content determine the relationship of insulin resistance with hepatic OXPHOS capacity in obesity. J Hepatol. 2025 Mar;82(3):417-426. doi: 10.1016/j.jhep.2024.08.012. Epub 2024 Aug 31. PMID 39218222
- [Derived] Sarabhai T, Kahl S, Gancheva S, Mastrototaro L, Dewidar B, Pesta D, Ratter-Rieck JM, Bobrov P, Jeruschke K, Esposito I, Schlensak M, Roden M. Loss of mitochondrial adaptation associates with deterioration of mitochondrial turnover and structure in metabolic dysfunction-associated steatotic liver disease. Metabolism. 2024 Feb;151:155762. doi: 10.1016/j.metabol.2023.155762. Epub 2023 Dec 19. PMID 38122893
- [Derived] Pafili K, Kahl S, Mastrototaro L, Strassburger K, Pesta D, Herder C, Putzer J, Dewidar B, Hendlinger M, Granata C, Saatmann N, Yavas A, Gancheva S, Heilmann G, Esposito I, Schlensak M, Roden M. Mitochondrial respiration is decreased in visceral but not subcutaneous adipose tissue in obese individuals with fatty liver disease. J Hepatol. 2022 Dec;77(6):1504-1514. doi: 10.1016/j.jhep.2022.08.010. Epub 2022 Aug 19. PMID 35988689
- [Derived] Apostolopoulou M, Gordillo R, Koliaki C, Gancheva S, Jelenik T, De Filippo E, Herder C, Markgraf D, Jankowiak F, Esposito I, Schlensak M, Scherer PE, Roden M. Specific Hepatic Sphingolipids Relate to Insulin Resistance, Oxidative Stress, and Inflammation in Nonalcoholic Steatohepatitis. Diabetes Care. 2018 Jun;41(6):1235-1243. doi: 10.2337/dc17-1318. Epub 2018 Mar 30. PMID 29602794
- See also: Homepage — https://ddz.de/studien/baria-ddz-studie/